CLINICAL TRIAL: NCT00737230
Title: Effective Management of Radiation-induced Bowel Injury: A Randomized Controlled Trial
Brief Title: Care of Cancer Patients With Bowel Injury Caused by Radiation Therapy to the Pelvis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Health Services Research
Other Study IDs: CDR0000601214; RMNHS-CCR2918-ORBIT; EU-20868
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Cancer
Keywords: long-term effects secondary to cancer therapy in adults; long-term effects secondary to cancer therapy in children; gastrointestinal complications; radiation toxicity; prostate cancer; bladder cancer; vulvar cancer; vaginal cancer; cervical cancer; endometrial cancer; anal cancer; rectal cancer; malignant testicular germ cell tumor
MeSH Terms: conditions — Neoplasms; Radiation Injuries; Prostatic Neoplasms; Urinary Bladder Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Anus Neoplasms; Rectal Neoplasms; Testicular Neoplasms | interventions — Early Intervention, Educational

INTERVENTIONS:
Other: educational intervention
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: gastrointestinal complications management/prevention
Procedure: management of therapy complications
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: A step-by-step procedure may help health care practitioners diagnose and treat cancer patients with bowel injury symptoms caused by radiation therapy.

PURPOSE: This randomized clinical trial is studying the care of cancer patients with bowel injury caused by radiation therapy to the pelvis.

DETAILED DESCRIPTION:
OBJECTIVES:

* To undertake a systematic review of the published effectiveness of investigations and treatments for patients with radiation-induced bowel injury after pelvic radiotherapy for cancer.
* To develop a diagnostic and treatment algorithm (based on evidence [where available] or on expert opinion [where there is no evidence]) for these patients.
* To examine each test in the algorithm for its usefulness in establishing precise diagnoses for these patients within the context of a randomized clinical trial.
* To examine whether use of the treatment algorithm in delivering treatment specifically targeted for each diagnosis improves symptoms and quality of life of these patients.
* To investigate whether the same level of care can be delivered to these patients by a nurse practitioner or by a specialist consultant gastroenterologist following the same algorithm.
* To identify other symptoms and healthcare needs experienced by these patients after pelvic radiotherapy and whether there are any other unmet needs in addition to their bowel injury.
* To determine the cost-effectiveness of the investigations and treatments developed for these patients.

OUTLINE: This is a two-part, multicenter study.

* Part 1: Researchers develop a diagnostic and treatment algorithm to guide health care practitioners in the management of patients with radiation-induced bowel injury. The algorithm, which is based on a systematic literature review or expert opinion, uses a series of simple tests to establish specific diagnoses and to target treatment for managing patient symptoms.
* Part 2: Patients are stratified according to tumor site (urological vs gynecological vs gastrointestinal) and degree of bowel dysfunction as measured by IBDQ-B score > 10 points above normal [< 60 vs 60-70]). Patients are randomized to 1 of 3 intervention arms.

  * Arm I (usual care): Patients receive an advice booklet on self-management of bowel symptoms. Patients whose symptoms continue 6 months after study enrollment may cross over to arm II.
  * Arm II: Patients undergo diagnostic and treatment algorithm-led management of bowel symptoms by a gastroenterologist.
  * Arm III: Patients undergo diagnostic and treatment algorithm-led management of bowel symptoms by a nurse practitioner.

Patients complete questionnaires about bowel symptoms and other pelvic symptoms, quality of life, and anxiety and depression at baseline, 6 months, and 1 year. Patients also complete questionnaires about cost effectiveness of the diagnostic and treatment algorithm or usual care.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Has undergone radical pelvic radiotherapy with curative intent to the prostate, bladder, vulva, vagina, cervix, endometrium, anus, or rectum OR para-aortic irradiation for a tumor at any of these primary sites, including the testes, > 6 months ago
* Has new-onset, troublesome gastrointestinal symptoms that developed > 6 months after completion of pelvic radiotherapy

  * Does not require immediate gastroenterological assessment, as deemed by the clinical oncologist
* Recruited directly from radiotherapy follow-up clinics at the Royal Marsden Hospital

PATIENT CHARACTERISTICS:

* Life expectancy > 1 year

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Improvement in gastrointestinal symptoms as measured by the modified IBDQ-B score, Rockwood Fecal Incontinence Quality of Life score, St Mark's Incontinence score, and the LENTSOMA score at baseline, 6 months, and 1 year

SECONDARY OUTCOMES:
Quality of life as measured by the modified IBDQ and SF-12 questionnaires at baseline, 6 months, and 1 year
Anxiety and depression scores as measured by the Hospital Anxiety and Depression Scale questionnaire at baseline, 6 months, and 1 year
Other pelvic symptoms (i.e., urinary function as measured by the ICSmaleSF and BFLUTSQ and sexual function as measured by the IIEF-6, ICSsex, and Jensen questionnaires) at baseline, 6 months, and 1 year
Cost-effectiveness of diagnostic tests and treatment compared to "usual care" as measured by the ED-5D questionnaire at 6 months and 1 year
Cost-effectiveness of nurse practitioner delivery of algorithm compared to gastroenterologist as measured by the ED-5D questionnaire at 6 months and 1 year
Other unmet healthcare needs as a direct result of pelvic radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jervoise Andreyev, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - London, London, England, United Kingdom

REFERENCES:
- [Derived] Andreyev HJ, Benton BE, Lalji A, Norton C, Mohammed K, Gage H, Pennert K, Lindsay JO. Algorithm-based management of patients with gastrointestinal symptoms in patients after pelvic radiation treatment (ORBIT): a randomised controlled trial. Lancet. 2013 Dec 21;382(9910):2084-92. doi: 10.1016/S0140-6736(13)61648-7. Epub 2013 Sep 23. PMID 24067488